CLINICAL TRIAL: NCT02474602
Title: Phototherapy Applied in Association of Muscle Training: Evaluation of Different Irradiation Protocols
Brief Title: Phototherapy Applied in Association With Strength Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Adriane Aver Vanin, MS, University of Nove de Julho
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Nove de Julho University; 2013/19355-3 (Other Grant/Funding Number: FAPESP-Brazil)
Record Dates: First submitted 2015-06-11; First posted 2015-06-18 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Muscle Development in Association to Phototherapy
Keywords: phototherapy; strength training; photobiostimulation; muscle development

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group A - Active or Placebo Phototherapy (Experimental): The phototherapy was divided in program 1 and program 2. One of these programs consisted in active phototherapy and the other placebo.
  The subjects allocated in group A, received program 1 before strength training, and the same program 1 after training.
  Interventions: Device: Active or Placebo Phototherapy (MR4)
- Group B - Active or Placebo Phototherapy (Experimental): The phototherapy was divided in program 1 and program 2. One of these programs consisted in active phototherapy and the other placebo.
  The subjects allocated in group B, received program 1 before strength training, and program 2 after training.
  Interventions: Device: Active or Placebo Phototherapy (MR4)
- Group C - Active or Placebo Phototherapy (Experimental): The phototherapy was divided in program 1 and program 2. One of these programs consisted in active phototherapy and the other placebo.
  The subjects allocated in group C, received program 2 before strength training, and program 1 after training.
  Interventions: Device: Active or Placebo Phototherapy (MR4)
- Group D - Active or Placebo Phototherapy' (Experimental): The phototherapy was divided in program 1 and program 2. One of these programs consisted in active phototherapy and the other placebo.
  The subjects allocated in group B, received program 2 before strength training, and the same program 2 after training.
  Interventions: Device: Active or Placebo Phototherapy (MR4)

INTERVENTIONS:
Device: Active or Placebo Phototherapy (MR4) — Participants performed a strength training. Forty-eight subjects practiced a training protocol with 80% of the load, measured through 1-repetition maximum test. The strength training lasted 12 weeks and the evaluations were done monthly. Phototherapy, active or placebo, were applied in 6 different points of quadriceps muscle depending the group randomized, before and after each training session.
  Other Names: MR4 device - device that combines super-pulsed lasers, and red and infrared LEDs (Multi Radiance Medical, Solon, OH, USA)

SUMMARY:
The effects of phototherapy has been widely studied by some research groups. The investigators know that there are positive results with light application to improve muscle performance and delay fatigue. However, there are few studies showing its´ effects on muscular training. Therefore, the aim of this study was to assess the effects of phototherapy applied at different times during 12 weeks of strength training. For such, 48 volunteers, healthy male, from 18 to 35 years old were recruited to perform a strength training protocol for the anterior muscle of the thigh development. Volunteers performed the training protocol twice a week for 12 weeks. There were assessed isometric peak torque in isokinetic dynamometer, 1-repetition maximum test in the leg extension and leg press machines and bilateral thigh perimetry.

DETAILED DESCRIPTION:
This is a clinical, randomized, controlled placebo and double-blind study. Forty-eight participants performed strength training protocol. Subjects practiced a protocol training with 80% of the load, measured through 1-repetition maximum test. The training protocol consisted in performing 5 sets of 10 repetitions, twice a week, employing leg extension and leg press machines.

Phototherapy, active or placebo, were applied in 6 different points of anterior muscle of the thigh before and after each training session. Only one investigator, that did not participate in any phase of the assessments and trainings sessions, knew about what program is active or placebo in phototherapy device. Randomisation carried out by a simple drawing of lots (A, B, C, or D) in the first visit. The phototherapy unit emitted the same sound regardless of the program used, active or placebo. Either strength training lasted 12 weeks and assessments were performed at baseline, 4, 8 and 12 weeks. There were evaluated maximal voluntary contraction (MVC), bilateral thigh perimetry and 1-repetition maximum test (1-RM).

ELIGIBILITY:
Inclusion Criteria:

There were included in the study

* healthy individuals,
* active,
* aged between 18 and 35 years old,
* male,
* presenting no history of musculoskeletal injury in the regions of the hip and knee in the two months prior to the study.
* that are not making use of pharmacological agents and / or nutritional supplements, and
* that have at least 80% of attendance to training.

Exclusion Criteria:

The participants were excluded if they

* present some musculoskeletal injury during the study

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2014-06; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Maximum voluntary contraction in the isokinetic dynamometer (MVC) | 12 weeks
  Functional performance measure

SECONDARY OUTCOMES:
1-Repetition Maximum test in the leg press and leg extension machines (1-RM) | 12 weeks
  Functional performance measure
Thigh perimetry | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto Cesar P Leal Junior, PhD, Study Director — University of Nove de Julho
Locations (1):
- Nove de Julho University, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Leal-Junior EC, Vanin AA, Miranda EF, de Carvalho Pde T, Dal Corso S, Bjordal JM. Effect of phototherapy (low-level laser therapy and light-emitting diode therapy) on exercise performance and markers of exercise recovery: a systematic review with meta-analysis. Lasers Med Sci. 2015 Feb;30(2):925-39. doi: 10.1007/s10103-013-1465-4. Epub 2013 Nov 19. PMID 24249354
- [Result] Seynnes OR, de Boer M, Narici MV. Early skeletal muscle hypertrophy and architectural changes in response to high-intensity resistance training. J Appl Physiol (1985). 2007 Jan;102(1):368-73. doi: 10.1152/japplphysiol.00789.2006. Epub 2006 Oct 19. PMID 17053104
- [Result] Antonialli FC, De Marchi T, Tomazoni SS, Vanin AA, dos Santos Grandinetti V, de Paiva PR, Pinto HD, Miranda EF, de Tarso Camillo de Carvalho P, Leal-Junior EC. Phototherapy in skeletal muscle performance and recovery after exercise: effect of combination of super-pulsed laser and light-emitting diodes. Lasers Med Sci. 2014 Nov;29(6):1967-76. doi: 10.1007/s10103-014-1611-7. Epub 2014 Jun 19. PMID 24942380